CLINICAL TRIAL: NCT02510326
Title: Evaluation of Motion in the Arthritic Wrist Joint
Status: Completed | Type: Observational
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Dr. Ronit Wollstein, Director hand and upper extremity service, Clalit Health Services
Other Study IDs: STT
Record Dates: First submitted 2014-03-23; First posted 2015-07-29 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Wrist Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The scaphotrapeziotrapezoid (STT) joint is a dome shaped joint in the radial wrist that is important in transfer of load from the thumb and radial hand to the scaphoid and the radioscaphoid and scaphocapitate joints. Arthritis in this joint is the second most common degenerative arthritis in the wrist, reported in 15% of wrist radiographs. The true incidence of arthritis in the STT joint however is unknown though we assume that most cases of arthritis are not clinically significant. Furthermore, the clinical and biomechanical significance of arthritis in this joint is unclear. The investigators' clinical impression is that the incidence of STT joint arthritis is inversely related to that of radiocarpal joint arthritis. In an ongoing study, we are examining the relationship between STT joint arthritis and radiocarpal joint arthritis on radiographs.

We suggest that STT joint arthritis alters the biomechanics of the wrist by limiting movement of the scaphoid within the STT joint thereby protecting the wrist from radiocarpal arthritis by limiting instability of the scaphoid.

The specific aims of this pilot study are to evaluate the movement of the arthritic scaphoid within the STT joint using a computer-generated model based on CT scan of the wrist and to compare this model with the already established model of the normal STT joint.

The investigators' hypothesis is that there is significantly less motion in the arthritic STT joint.

DETAILED DESCRIPTION:
Because it is poorly understood, the treatment of wrist arthritis remains limited to suboptimal salvage operations and wrist fusions. These are surgeries, which greatly limit function. This study is designed to evaluate arthritis of the STT joint and its affect on arthritis in other parts of the wrist. This may improve the understanding of wrist mechanics enabling us to develop better treatment of wrist arthritis. STT joint arthrodesis is an accepted surgery whose indications may be influenced by information obtained in this study.

Five patients being treated by the PI that have a diagnosis or a finding of STT joint arthritis stage 3 on X-ray will be included in the study. The radiographs are standard of care for various hand and wrist conditions and patients will be sent for radiographs only as part of their care. The patients will be eligible for the study following informed consent. The CT scan will be performed at 5-7 wrist positions: neutral, maximum extension, flexion, radial deviation, ulnar deviation (plus radial extension and ulnar flexion for 7 positions). Slice thickness will be less than 1 mm. The slices will be located between distal radioulnar joint (DRUJ) and the 2nd carpometacarpal (CMC) joint. The CT scans will then be sent for evaluation by the computer based kinematic program. No identifiable information will be collected or recorded. The program will develop a kinematic model of the STT joint in the presence of arthritis.

The model (kinematic data) will be compared to an existent "normal" model, based on 7 CT scans of normal STT joints. This data is already in existence and therefore no normal wrists are accrued.

ELIGIBILITY:
Inclusion Criteria:

Patients with STT joint osteoarthritis(OA) - stage 3

Exclusion Criteria: incomplete radiographs, early stage STT OA

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Five patients being treated by the PI that have a diagnosis or a finding of STT joint arthritis stage 3 on X-ray will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
motion in the STT joint | 1 year
  A kinematic model based on data from the wrist CT acquired in the different wrist positions.(kinematic data) will be compared to an existent "normal" model, based on 7 CT scans of normal STT joints.

CONTACTS AND LOCATIONS:
Locations (1):
- Carmel Medical Center, Haifa, Israel